CLINICAL TRIAL: NCT00893009
Title: The Effect on Small Airways of Addition of Theophylline as Inducer of Histone Deacilase Activity for Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD), Treated With Inhaled Steroids and Long Acting Beta Agonists
Acronym: COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: David Stav MD, Pulmonary Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02/09
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2009-04

CONDITIONS: COPD
Keywords: Forced expiratory volume in one second; Inspiratory capacity; endurance time; residual volume
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Theophylline (Active Comparator): 100 twice a day
  Interventions: Drug: Theophylline

INTERVENTIONS:
Drug: Theophylline — 100 mg twice a day
  Arms: Theophylline
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic progressive respiratory disorder causing disability with an increasing burden to the patient, his family and to the health services. Treatment of COPD patients depends on the stage of the disease. COPD responds poorly to corticosteroids, in spite of inflammation is a major component in its pathogenesis. A major barrier to therapy of COPD is resistance to the anti-inflammatory effects of corticosteroids. The molecular mechanisms for this corticosteroid resistance are now being elucidated, particularly as the molecular basis for the anti-inflammatory effects of corticosteroids is better understood (12). An important mechanism of corticosteroid resistance in COPD, which is also linked to amplification of the inflammatory process, is a reduction in the critical nuclear enzyme histone deacetylase (HDAC)2 . Since the major changes are at the level of small airways. We will examine the effect of addition of theophylline product to stable COPD patients treated with combined inhaler of inhaled corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* stable stage II and III (GOLD) COPD, diagnosed 2 years ago and up

Exclusion Criteria:

* Heart failure Malignancy Immune suppressed

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Air trapping | 1 year

SECONDARY OUTCOMES:
endurance time | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonar Institute, Assaf Harofeh Medical Center, Beer Yaakov, Israel